CLINICAL TRIAL: NCT02552784
Title: Determinants of Health Status and Quality of Life of Patients and Their Parents With Inherited Metabolic Diseases Diagnosed During Childhood and Requiring Restrictive and Specific Diet
Brief Title: Quality of Life of Patients and Theirs Parents With Inherited Metabolic Diseases With Restricted Diet
Acronym: MHMRSQol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-38; 2014-A01874-43 (Registry Identifier: Ansm)
Record Dates: First submitted 2015-07-01; First posted 2015-09-17 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Inherited Metabolic Diseases Requiring Restrictive and Specific Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- patients and their parents with inherited metabolic diseases (Experimental): The population is a dynamic/open cohort consists of all patients MHMRS diagnosed and supported in one of the six Centers of Reference for Metabolical disease or one of the three Centers of Competence for Hereditary Metabolic Diseases or in the Center of Réference for Hereditary liver Metabolism Diseases since 2000. For each patient, the date of entry into the cohort is the diagnostic date of MHMRS. The study includes all prevalent and incident cases .
  Interventions: Behavioral: data assessment of the state of health and quality of life of patients and their families

INTERVENTIONS:
Behavioral: data assessment of the state of health and quality of life of patients and their families — Study medical determinants, socioeconomic, behavioral, environmental of health, school and professional integration, and short- and medium-term quality of life of all patients residing in France for which the diagnosis of hereditary diseases metabolism with specific diet (MHMRS) was performed during their childhood.

SUMMARY:
The general objective is study medical, socioeconomic, behavioral, health environmental, school and professional integration, and short- and medium- term quality of life determinants for all patients under 18 years old, residing in France for which the diagnosis of inherited metabolic diseases with specific regime (MHMRS) has been achieved during their childhood.

DETAILED DESCRIPTION:
The study population is a dynamic/open cohort consists of all patients MHMRS diagnosed and supported in one of the six Centers of Reference for Metabolical disease or one of the three Centers of Competence for Hereditary Metabolic Diseases or in the Center of Réference for Hereditary liver Metabolism Diseases since 2000. For each patient, the date of entry into the cohort is the diagnostic date of MHMRS. The study includes all prevalent and incident cases .

The evaluations include all data collected by querying patients and their families and medical data collected by the medical team.

The data collected concern in one hand explanatory variables characterizing the state of health and quality of life of patients, on the other variables describing the factors considered as potential determinants, namely:

* Socio -demographic and socio-economic on the patient and family.
* Clinical and therapeutic relative to the patient : age at the time of diagnosis, illness and consequences, type of treatment and diet.
* On possible alterations of physical health: overall assessment of the importance of using health professionals and specific description of the various physical health problems.
* Psycho- behavioral and cognitive.
* Quality of life of patients and their family.
* On the patient's relationship with the care system (access to care and satisfaction).

The frequency of evaluations is 2 years. The evaluation will be at a consultation in the usual medical monitoring way up conducted in these children, allowing to collect clinical information directly nearby medical teams that support them.

The various measurement tools used are:

* STAI-C and STAI-Y
* BRIEFCOPE and KIDCOPE
* GOODMAN questionnaire
* FAS questionnaire
* WECHSLER scale
* VSPA, VSPA-e and VSPA-p
* QUALIN
* WHOQOL-BREF

The project is under the authority of a Steering Committee comprising representatives of all the partners in the project teams. The project is supervised by the Scientific Council of the SFEIM (Société Francaise pour les Erreurs Inées du Métabolisme) and the G2M (Groupement des centres de référence et de compétence des Maladies héréditaires du Métabolisme) which is consulted on the scientific guidance of the project.

At the end of a study report will be prepared. It will detail all the decisions inherent in the conduct of the project and the results obtained. This report will be sent to the Ministry of Health under the cover of the Delegation for Clinical Research. The report will form the basis of the adjacent communications will be co-signed by the members of the Steering Committee and will reference the origin of the aid received.

ELIGIBILITY:
Inclusion Criteria:

Included in MHMRS databases from different centers

* Age less than 18 years at diagnosis
* Diagnostic MHMRS made from 01/01/2000
* Treatment and management of MHMRS initiated in one of the clinical sites
* Living in France

  * Living
  * Compliance with criteria for inclusion in the cohort
  * Having agreed to participate in the study
  * Allowed to participate in the study by the parents or legal guardians for any minor subject.

Exclusion Criteria:

* Can't be included subjects not complying with at least one of the inclusion criteria previously mentioned .
* Excludes all subjects at least one of the following criteria:

  * Moving outside France after baseline ( initial treatment performed in one of the participating centers )
  * Withdrawal of consent / refusal of monitoring;
  * Not responding at three successive waves of investigation.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 763 (Estimated)
Dates: Start 2015-01; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient's anxiety assessment | 6 years
  Anxiety assessment of children by autoquestionnaires: STAI-C (8-10 years old); STAI-Y (11-17 years old); STAI (patients becoming adults)
Assessment of adaptive coping strategies of patients | 6 years
  Assessment of adaptive coping strategies of patients by questionnaires (BriefCope for adults patients, Kidcope for young patients)
Patient's behavior assessment | 6 years
  Assessment of child's behavior by Strengths and difficulties questionnaires and assessment of adult's behavior by the sociale adaptation scale (Weintraub scale)
Patient's quality of life assessment | 6 years
  Patient's quality of life assessment by VSP-A questionnaire
Parent's quality of life assessment | 6 years
  Parent's quality of life assessment by WHOQOL-BREF questionnaire
Assessment of adaptive coping strategies of parents | 6 years
  Assessment of adaptive coping strategies of parents by BriefCope questionnaire
Parent's anxiety assessment | 6 years
  Parent's anxiety assessment by STAI questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Hôpital de la Timone Assistance Publique Hôpitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Ouattara A, Resseguier N, Cano A, De Lonlay P, Arnoux JB, Brassier A, Schiff M, Pichard S, Fabre A, Hoebeke C, Guffon N, Fouilhoux A, Broue P, Touati G, Dobbelaere D, Mention K, Labarthe F, Tardieu M, De Parscau L, Feillet F, Bonnemains C, Kuster A, Labrune P, Barth M, Damaj L, Lamireau D, Berbis J, Auquier P, Chabrol B. Individual and Family Determinants for Quality of Life in Parents of Children with Inborn Errors of Metabolism Requiring a Restricted Diet: A Multilevel Analysis Approach. J Pediatr. 2023 Mar;254:39-47.e4. doi: 10.1016/j.jpeds.2022.08.060. Epub 2022 Oct 17. PMID 36265570